CLINICAL TRIAL: NCT03416608
Title: Patient Experiences of Use of Point-of-Care Ultrasound in General Practice: A Questionnaire Study
Brief Title: Patient Experiences of Use of Point-of-Care Ultrasound in General Practice
Status: Completed | Type: Observational
Sponsor: Aalborg University (Other)
Responsible Party: Principal Investigator, Camilla Aakjær Andersen, Principal Investigator, Aalborg University
Other Study IDs: GULD-patient questionnaire
Record Dates: First submitted 2018-01-10; First posted 2018-01-31 (Actual); Last update posted 2018-12-12 (Actual); Status verified 2018-12

CONDITIONS: Ultrasound; General Practice
Keywords: ultrasound; patient experience; diagnostic test; general practice; family medicine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study in part of a larger cohort study (clinical trials ID number: NCT03375333) that examine the use of ultrasound in general practice.

In the present study patient experiences, with use of ultrasound in the consultation at the general practitioners office, will be explored through a questionnaire.

DETAILED DESCRIPTION:
This study is a Cross-sectional study, which is conducted as part of a larger cohort study: How Point-of-Care Ultrasound (POC-US) Affects the Diagnostic Process in General Practice. A prospective follow-up study. (Clinical trials registration number: NCT03375333)

Study setting:

The study will take place in 20 different general practices in Denmark where the general practitioners (GPs) use POC-US.

Interventions There is no intervention in this study. The registration in this study will reflect GPs routine daily use of POC-US not adding more examinations or in other ways influence on the treatment of patients.

Sample size Twenty general practitioners (GPs) are expected to use POC-US 2-3 times a day, and assuming a participation rate of 80%, there will be between 640-960 US scan during the study period of one month.

Recruitment All patients who consult the participating GP for conditions relevant for a POC-US examination will be offered to participate in the study. Patients are excluded if they do not wish to participate or if they are not able to give an informed consent.

Patients must provide written, informed consent before any study procedures occur. Only patients assigned to the GPs practice can participate in the study.

Data collection method After the consultation in the GP's office, patients will be asked to fill out a questionnaire about their experience with POC-US in the consultation. The GPs will provide the patients with a unique ID-number and a link to an online questionnaire on the SurveyXact server. The patients will access the online questionnaire using this ID-number through Ipads or on a paper edition.

Baseline information regarding the participating GPs will be provided through the original study. Baseline questions about the patients will be part of the patient-questionnaire following the consultation.

The items in this questionnaire are generated from a qualitative interview study with GPs working in general practice and using POC-US. The items are the GPs expressed believes and concerns about how ultrasound was experienced by their patients.

This questionnaire is developed through the following steps:

1. A first edition of the questionnaire is developed based on the results of a qualitative interview study with Danish GPs on their experiences on how ultrasound can be used in general practice.
2. To test face validity, comprehension and wording of the questionnaire, pilot tests are done with laypeople and patients,using the "think-aloud" technique and cognitive interviewing. The pilot-tests are done in two geographical-separated clinics including five patients in each clinic. Adaptions and rephrasing follow after the results are compared.
3. A validation test will include presenting the rephrased questions from the pilot-tests to 5 GPs, who use ultrasound, and asking them to compare the phrased questions to the original items from the qualitative interviews. Adaptions will follow.
4. A final pilot-test will include interviews with patients, who have been ultrasound scanned in two other clinics using the "Think-aloud" technique. In this pilot-test the patients are presented to both a paper-version and an online-version of the questionnaire, to test functionality and feasibility. Pilot-tests and adaptions will continue until the questionnaire is completed without difficulties.

Retention Participant Retention GPs will be asked to register not-included patients, in whom POC-US was used during the study period, on a separate form and to declare the reason for the failed inclusion of the patient.

Participant Withdrawal Participating GPs and patients may withdraw from the study for any reason at any time.

Data management Data will be saved electronically in the SurveyXact server and on a server at Aalborg University and will only be accessed by the research group using passwords.

The Research Unit for General Practice in Aalborg is the Data Controller. Each participating GP will be data processor and can only process data pursuant to an agreement with the data controller. A data processor agreements will be made between the Research Unit for General Practice in Aalborg and each participating GP, between the Research Unit for General Practice in Aalborg and Aalborg University, and between Aalborg University and SurveyXact according to the Danish Data Protection Agency recommendations.

The Key files identifying the patients will be safely stored at the GPs office and the research group will not have access to this information during the study.

Statistics The questionnaire data will be collected on an ordinal scale and reported descriptively using frequencies. The correlation between the GPs reported confidence in the tentative diagnosis on a numeric rating scale from 1-5 perceived at an ordinal scale and patients reported experience of ultrasound in the consultation will be compared using scatterplots and Goodman and Kruskal's gamma will be used to test association.

Data monitoring During the study period the research team will be able to observe if the GPs include patients in the study and make contact to the GPs who fail to include patients in order to help out with any difficulties.

Harms All adverse events occurring during the study will be registered.

Research ethics approval The studies are approved by the Danish Data Protection Agency and the Committee of Multipractice Studies in General Practice in Denmark.

Consent or assent Prior to participation, patients will receive written and oral information and a written consent to participate will be obtained.

If a GP or a patient wished to redraw their consent to participate in the study, the GP will contact the research team and no further data will be collected.

Protocol amendments Will be declared and all editions and changes in the protocol will be saved.

Confidentiality All participating GPs have signed a confidentiality agreement.

Declaration of interest None

Access to data Only the Research team will have access to data.

ELIGIBILITY:
Inclusion criteria:

- All patients, who the GP intends to examine with POC-US.

Exclusions criteria:

* Patient not willing or able to give informed consent
* Patients previously included in the study

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study will take place in 20 different general practices in Denmark where the GPs use POC-US. The participating GPs will try to include all patients were they use POC-US in the consultation.
  Patients must provide written, informed consent before any study procedures occur (see Appendix 1 for sample Informed Consent Form). Only patients assigned to the GPs practice can participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 579 (Actual)
Dates: Start 2018-01-15 (Actual); Primary Completion 2018-09-01 (Actual); Study Completion 2018-09-02 (Actual)

PRIMARY OUTCOMES:
Information | assessed immediately after the ultrasound examination
  This domain will be explored through the following questions:
  Were you informed about the purpose of the ultrasound examination? Were you informed about the difference between a specialist ultrasound and a GP ultrasound? Were you informed about the result of the ultrasound examination?
Influence on the consultation | assessed immediately after the ultrasound examination
  This domain will be explored through the following questions:
  Did you think the ultrasound examination was a natural part of the consultation? Did you think the ultrasound examination was disruptive in the consultation? Did the ultrasound examination influence the relationship between the GP and you? Do you think ultrasound made a difference in the consultation?
Diagnostic reassurance | assessed immediately after the ultrasound examination
  This domain will be explored through the following questions:
  Do you feel more thoroughly examined after the ultrasound examination? Do you have a better understanding of your health problem after the ultrasound examination? Do you feel more at ease after the ultrasound examination? Has your confidence in the GPs diagnosis changed after the ultrasound examination? Has the ultrasound examination changed your feeling of being taken seriously?
Patient satisfaction | assessed immediately after the ultrasound examination
  This domain will be explored through the following questions:
  Was your overall experience with ultrasound in the GP's office positive or negative? Would you recommend ultrasound in the GPs office to others? Do you think ultrasound is a service improvement in the GP's office? Do you think ultrasound is a quality improvement in the GP's office?

SECONDARY OUTCOMES:
Associations between GP confidence in the diagnosis and patients sense of diagnostic reassurance | assessed immediately after the ultrasound examination
  Association between GPs declared confidence in the tentative diagnosis after using ultrasound in the consultation (data from the original cohort expressed on a scale from increased confidence to decreased confidence) and patients' answers to the question "Has your confidence in the GPs diagnosis changed after the ultrasound examination?" expressed on a scale from decreased to increased confidence.
Associations between GP confidence in the diagnosis and patients experience of improved care | assessed immediately after the ultrasound examination
  Association between GPs declared confidence in the tentative diagnosis after using ultrasound in the consultation (expressed in the original cohort on a scale from increased confidence to decreased confidence) and patients' answers to the question "Do you feel more at ease after the ultrasound examination?" expressed on a scale from less at ease to more at ease.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Bach Jensen, Professor, GP, PhD, Study Chair — Aalborg University
Locations (1):
- Research unit for general practice in Aalborg,department of clinical medicine Aalborg university, Aalborg, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Andersen CA, Brodersen J, Rudbaek TR, Jensen MB. Patients' experiences of the use of point-of-care ultrasound in general practice - a cross-sectional study. BMC Fam Pract. 2021 Jun 18;22(1):116. doi: 10.1186/s12875-021-01459-z. PMID 34144701

DOCUMENTS (1):
  • Study Protocol (2018-01-29): https://cdn.clinicaltrials.gov/large-docs/08/NCT03416608/Prot_000.pdf